CLINICAL TRIAL: NCT06372275
Title: Reframing Health Behavior Change: A Randomized Controlled Trial of a Relational Frame Theory (RFT)-Informed Values Intervention for Health
Brief Title: Investigating Two Prototype Mobile App Interventions to Increase Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mississippi State University (Other)
Collaborators: Association for contextual behavioral science (Unknown)
Responsible Party: Principal Investigator, Jennifer Krafft, Assistant Professor, Mississippi State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2024-03-28; First posted 2024-04-17 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Health-Related Behavior
Keywords: Physical Activity; Exercise; Values Clarification; Self-Reflection; Acceptance and Commitment Therapy; Mobile App; Motivation
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Values Clarification Condition (Experimental): Participants will respond to values clarification writing prompts related to physical exercise once a day over 28 days in addition to a short daily survey. In each session, one writing prompt will be randomly presented from a pool of four categories: hierarchical, conditional, distinction, and perspective-taking. The survey inquires about time spent doing light, moderate, and vigorous exercise the day before, in addition to time spent watching television, using the computer, and sitting. It also includes the 24 item Multidimensional Psychological Flexibility Inventory adapted for ecological momentary assessment and questions asking participants to rate the extent to which they currently feel 8 emotions, their current motivation to exercise, and their stress yesterday. The writing prompt and survey are estimated to take 10 minutes to complete daily. Participants will have the option to review additional educational content about values and their previous written responses.
  Interventions: Behavioral: Values Clarification Mobile Application
- Self-Reflection Condition (Placebo Comparator): Participants in this condition will be asked to respond to one randomly selected self-reflection prompt about physical activity from a library of 28 prompts once a day over 28 days [4 weeks]. As with the experimental condition, participants will also complete the same daily survey which includes questions about how many minutes they spent doing light, moderate, and vigorous exercise the day before, in addition to how many hours they spent watching television, using the computer, and sitting. The survey also contains the 24 item Multidimensional Psychological Flexibility Inventory adapted for ecological momentary assessment and questions asking participants to rate the extent to which they are currently feeling 8 emotions, their current motivation to exercise, and their stress the day before. This is estimated to take 10 minutes to complete daily. Participants will have the option to review additional educational content about values clarification and their previous written responses.
  Interventions: Behavioral: Self-Reflection Mobile Application

INTERVENTIONS:
Behavioral: Values Clarification Mobile Application — Participants in the intervention group will be asked to answer a series of values clarification writing prompts related to physical activity once a day over four weeks.
  Arms: Values Clarification Condition
Behavioral: Self-Reflection Mobile Application — Participants in the control group will be administered writing prompts in the same format and frequency as the values intervention, but with prompts focused on self-reflection related to physical activity.
  Arms: Self-Reflection Condition

SUMMARY:
This randomized control trial aims to investigate whether writing about personal values helps enhance motivation to engage in physical activity, relative to general self-reflective writing. This study will help to (1) assess whether values clarification leads to increased motivation to engage in physical activity, greater stability in motivation, and improvements in engagement in physical activity and valued action, relative to engaging in self-reflection, (2) determine if the impact of values clarification on these outcomes vary depending on context (e.g., positive/negative affect, psychological inflexibility, stressful events), (3) explore whether values clarification procedures that employ distinct relational frames (hierarchical, conditional, distinction, and deictic) differentially impact motivation to engage in physical activity, and daily engagement in physical activity, and (4) explore whether the impact of values clarification vary depending on baseline self-compassion and/or intrinsic/extrinsic motivation.

DETAILED DESCRIPTION:
This randomized control trial study aims to investigate the efficacy of a values clarification prototype mobile application intervention in increasing physical activity and enhancing motivation to exercise in a general, adult sample. Participants will be recruited using a variety of recruitment methods (e.g., Google Ads, posts on relevant online groups such as Facebook groups, posting flyers, and provider referrals). Interested participants will first complete an online pre-screening asking whether they are between the ages of 18 and 65, reside in the United States, want to increase their physical activity, own a device that can receive text messages, and have reliable internet access. Participants will also be asked about why they want to participate in the study, about their current level of physical activity and how they hope to change it, and about how they learned about the study. Those who meet the eligibility criteria in the pre-screening will be directed to review an online informed consent form. Those who indicate that they consent will be directed to provide their contact information (name, email, and phone number). A trained research assistant will call the participant to ask additional screening questions assessing all exclusion criteria (listed later in this registration). Eligible participants at this stage will be redirected to complete a baseline survey and then be randomly assigned to either the: (1) Experimental group with the values clarification mobile application or (2) the control group with the self-reflection mobile application. Participants will have access to the app hosted on Qualtrics for 28 days. They will first complete a tutorial, and then begin completing the daily surveys in addition to the writing prompts. Participants will receive daily text message reminders to use the app at a time that they specify. Four weeks after baseline, participants will be asked to complete a post-treatment survey and eight weeks after baseline, participants will be asked to complete a final, follow-up survey. Participants will be given the opportunity to use the alternative app at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old.
2. Living in the United States
3. Own a device that can receive text messages.
4. Have reliable internet access.
5. Want to increase physical activity.

Exclusion Criteria:

1. Below 18 or above 65 years old.
2. Living outside the United States
3. Not owning a device that can receive text messages.
4. Not having reliable internet access.
5. Not interested in increasing physical activity.
6. Not having the fluency in English sufficient to read or understand study materials.
7. Unable to engage in physical activity safely due to medical status.
8. Currently in another program focused on increasing physical activity.
9. Currently taking medications that cause dizziness or feeling faint while standing (e.g. some hypertension medications).
10. Already completing 150 minutes or more of moderate-to-vigorous physical activity most weeks.
11. Report any condition that would preclude adherence to the intervention protocol (e.g. current or past substance use disorder or psychiatric hospitalization, terminal illness diagnosis.)
12. Participants will also be excluded from the study if they are suspected of being a bot or invalid respondent based on their responses.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) - Total physical activity | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures physical activity. The IPAQ comprises 27 items that assess time spent engaging in various levels of physical activity / time spent sitting and participants are asked to report their responses in terms of minutes, hours, or days. Scores can be computed continuously or categorically. Continuous scoring will be used. Total physical activity will be the primary outcome; components of physical activity and sedentary time will be examined as secondary outcomes. The investigators added an additional item at the end of the survey: "Was your physical activity much less than typical this week due to very unusual circumstances such as being sick, moving, unusual travel, being hospitalized, etc.?" Response options were: "Yes - my physical activity this week was much less than typical due to very unusual circumstances", "No - my physical activity was fairly typical despite experiencing very unusual circumstances", and "No - my circumstances were basically normal".

SECONDARY OUTCOMES:
Behavioral Regulation in Exercise Questionnaire, Version 3 (BREQ-3) - Total score | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures an individual's motivation to exercise according to self-determination theory (SDT). The BREQ-3 consists of 24 items that are rated on a scale from 0 (not true for me) to 4 (very true for me). Scores range from a minimum of 0.0 to a maximum of 4.0 for each motivation type, with higher scores indicating a greater level of endorsement of the specific motivation dimension. A global score called the Relative Autonomy Index can be calculated.
Amotivation - Subscale of the Behavioral Regulation in Exercise Questionnaire, Version 3 (BREQ-3) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Amotivation" subscale of the BREQ-3 refers to a non-self-determined form of regulation, where there is no intention at all to engage in exercise. A sample item is "I don't see why I should have to exercise."
External Regulation - Subscale of the Behavioral Regulation in Exercise Questionnaire, Version 3 (BREQ-3) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "External Regulation" subscale of the BREQ-3 refers to motivation that is externally regulated by compliance, conformity, or external rewards and punishment and that is not self-determined. A sample item is "I exercise because other people say I should."
Introjected Regulation - Subscale of the Behavioral Regulation in Exercise Questionnaire, Version 3 (BREQ-3) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Introjected Regulation" subscale of the BREQ-3 refers to motivation that is driven by self-control, an effort to maintain self-esteem, and/or internal rewards and punishments. A sample item is "I feel guilty when I don't exercise."
Identified Regulation - Subscale of the Behavioral Regulation in Exercise Questionnaire, Version 3 (BREQ-3) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Identified Regulation" subscale of the BREQ-3 refers to motivation that is based on the conscious acceptance of exercise as a personal value that overrides any difficulties or obstacles in its way. A sample item is "I think it is important to make the effort to exercise regularly."
Integrated Regulation - Subscale of the Behavioral Regulation in Exercise Questionnaire, Version 3 (BREQ-3) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Integrated Regulation" subscale of the BREQ-3 refers to motivation to exercise that is fully congruent with one's identity. Integrated Regulation is fully self-determined since it is engaged in willingly. However, it is distinguished from intrinsic motivation because the reason behind engaging in the behavior (i.e., exercise) is still for separable outcomes and not for the sake of itself. A sample item is "I exercise because it is consistent with my life goals."
Intrinsic Regulation - Subscale of the Behavioral Regulation in Exercise Questionnaire, Version 3 (BREQ-3) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Intrinsic Regulation" subscale of the BREQ-3 refers to motivation to exercise that is entirely motivated by interest and enjoyment inherent in exercise itself. It is fully self-motivated and self-determined. A sample item is "I get pleasure and satisfaction from participating in exercise."
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Questionnaire v1.2 | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures an individual's general mental, physical, and social health. This scale consists of 10 items, 9 of which are rated on a scale from 1 (poor) to 5 (excellent), and 1 item pertaining to pain that is rated on a scale from 0 (no pain) to 10 (worst pain imaginable). Overall, higher scores indicate better global health. Scores can be calculated using either the HealthMeasures Scoring Service, which uses response pattern scoring, or by using the manual to convert raw scores to t-scores.
Global Mental Health - Subscale of the PROMIS Global Health Questionnaire v1.2 (Patient-Reported Outcomes Measurement Information System) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Global Mental Health" subscale of the PROMIS Global Health questionnaire v1.2 provides a generic self-assessment of one's mental health. A sample item is "In general, how would you rate your mental health, including your mood and ability to think?"
Global Physical Health - Subscale of the PROMIS Global Health Questionnaire v1.2 (Patient-Reported Outcomes Measurement Information System) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Global Physical Health" subscale of the PROMIS Global Health questionnaire v1.2 provides a generic self-assessment of one's physical health. A sample item is "In general, how would you rate your physical health?"
Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Satisfaction with Social Roles and Activities 8a | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures satisfaction with performing one's usual social roles and activities. The scale consists of 8 items that are rated on a scale from 1 (not at all) to 5 (very much). Scores can be calculated using either the Assessment Center Scoring Service, which uses response pattern scoring, or by using the manual to convert raw scores to t-scores. Higher scores indicate better satisfaction with one's social role and activities.
Multidimensional Psychological Flexibility Inventory - Short Form 24-item version (MPFI-24) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures psychological flexibility and psychological inflexibility. The scale consists of 24 items, and participants are asked to consider the past two weeks and select a response from a scale ranging from "Never True" to "ALWAYS True". A global score on psychological flexibility and inflexibility is produced, in addition to subscale scores pertaining to each of the six dimensions of psychological flexibility and inflexibility. Scores range from a minimum of 1.0 to 6.0, with higher scores reflecting higher levels of the domain being assessed (i.e., psychological flexibility or inflexibility, etc.).
Contact With Values - Subscale of the Multidimensional Psychological Flexibility Inventory - Short Form 24-item version (MPFI-24) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Contact With Values" subscale of the MPFI-24 falls under the psychological flexibility factor and measures the extent to which an individual is connected to what is important to them in life, giving direction to their actions. Participants are asked to consider the past two weeks when rating their responses, and a sample item is: "I was very in-touch with what is important to me and my life."
Lack of Contact With Values - Subscale of the Multidimensional Psychological Flexibility Inventory - Short Form 24-item version (MPFI-24) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  The "Lack of Contact With Values" subscale of the MPFI-24 falls under the psychological inflexibility factor and measures the extent to which an individual is disconnected from their values in their daily life. Participants are asked to consider the past two weeks when rating their responses, and a sample item is: "When life got hectic, I often lost touch with the things I value."
Values Clarity Questionnaire (VCQ) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures how well respondents understand and can articulate their values. The VCQ consists of 7 items rated on a scale from 1 (strongly disagree) to 5 (strongly agree). Total scores range from a minimum of 7 to a maximum of 35, with higher scores indicating higher levels of clarity, understanding, and articulation of one's own values.
Self-Compassion Scale Short Form (SCS-SF) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures global self-compassion across six factors: self-kindness, self-judgment, common humanity, isolation, and mindfulness. The SCS-SF consists of 12 items rated on a scale from 1 (almost never) to 5 (almost always). Total scores range from a minimum of 1.0 to a maximum of 5.0, with higher scores indicating greater levels of self-compassion.
Random responding question | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  Participants will be asked to choose one of the following statements that best describe their participation in the survey, noting that their answer does not impact their participation in the study in any way: "I answered every question carefully and honestly" (1); "I answered most questions carefully and honestly" (2); "I randomly responded and/or did not respond honestly to about half of the questions" (3); "I randomly responded and/or did not respond honestly to most questions" (4); and "I randomly responded and/or did not respond honestly to any questions" (5). Participants who score a 4 or 5 will be screened out for random responding.
Credibility & Expectancy Questionnaire (CEQ) | After the app tutorial (approximately 0-1 weeks after baseline)
  A self-report measure of the perceived credibility of and expectations toward a treatment. The CEQ consists of 6 items, 3 for Credibility and 3 for Expectancy. An average score ranging from 1 to 9 will be calculated for Credibility, with higher scores a greater perception of the intervention's credibility by the participants. For the expectancy component, an average percentage score will be calculated ranging from 0% to 100%, with higher percentages indicating more positive expectations towards the treatment.
System Usability Scale (SUS) | Posttreatment (4 weeks after baseline)
  A self-report measure of usability of a technological system. The SUS consists of 10 items rated on a scale from 1 (strongly disagree) to 5 (strongly agree). Scores are summed and doubled such that they range from 0 to 100 (as per the official scoring instructions), with high scores indicating greater usability.
Treatment Evaluation Inventory-Short Form (TEI-SF) | Posttreatment (4 weeks after baseline)
  A self-report measure of treatment acceptability. The TEI-SF consists of 7 items rated from 1 (strongly disagree) to 5 (strongly agree). Scores range from 7 to 35, with higher scores indicating higher levels of endorsement for treatment acceptability.
Exercise ecological momentary assessment (EMA) questions | Daily during 28 days of mobile prototype app intervention
  Participants are asked to respond to questions used in previous research that assess the time spent in the past 24 hours (in minutes) in moderate-intensity physical activity and vigorous-intensity physical activity, in addition to time spent (in hours) on sedentary time. Response options were modified to allow participant to enter minutes rather than selecting a category. The three questions assessing sedentary time asked about how many hours were spent watching television, using the computer, and sitting. The investigators included an additional question assessing light-intensity physical activity.
Multidimensional Psychological Flexibility Inventory - Short Form 24-item version adapted for ecological momentary assessment (MPFI-24 validated for EMA) | Daily during 28 days of mobile prototype app intervention]
  The MPFI-24 was adapted for ecological momentary assessment (EMA) purposes, making it a self-report scale that assesses momentary psychological flexibility and inflexibility. Participants are asked to consider their day yesterday and rate their responses on a scale ranging from "NEVER True" to "ALWAYS True". Scores range from a minimum of 1.0 to 6.0, with higher scores reflecting higher levels of the domain being assessed (i.e., momentary psychological flexibility or inflexibility, etc.).
Momentary Contact With Values - Subscale of the Multidimensional Psychological Flexibility Inventory - Short Form 24-item version adapted for ecological momentary assessment (MPFI-24 validated for EMA) | Daily during 28 days of mobile prototype app intervention]
  The "Contact With Values" subscale of the MPFI-4 adapted for EMA falls under the psychological flexibility factor and measures momentary connectedness to one's values. Participants will be asked to consider their experience the day before when rating their responses, and a sample item is: "I stuck to my deeper priorities in life."
Momentary Lack of Contact With Values - Subscale of the Multidimensional Psychological Flexibility Inventory - Short Form 24-item version adapted for ecological momentary assessment (MPFI-24 validated for EMA) | Daily during 28 days of mobile prototype app intervention]
  The "Lack of Contact With Values" subscale of the MPFI-4 adapted for EMA falls under the psychological inflexibility factor and measures the extent to which one is not connected to their values at the moment. Participants will be asked to consider their experience the day before when rating their responses, and a sample item is: "My priorities and values often fell by the wayside."
Emotion ratings | Daily during 28 days of mobile prototype app intervention
  Participants will be asked to rate the extent to which they feel 8 emotions in the present moment. The question is: "Rate how ___ you feel right now". The items are: "Content", "Relaxed", "Enthusiastic", "Joyful", "Anxious", "Angry", "Sad", and "Ashamed". The rating scale provided ranges from 1 (very slightly or not at all) to 5 (very much). As in past studies the investigators have conducted, the scale was adapted to replace "sluggish" with "ashamed."
Current Motivation to Exercise | Daily during 28 days of mobile prototype app intervention
  Participants will be asked about their current motivation level to exercise. The question is: "How motivated are you right now to exercise?" The rating scale provided ranges from 1 (not at all) to 7 (extremely). This question will be asked both before and after the writing exercise.
Previous Day Stress Level | Daily during 28 days of mobile prototype app intervention
  Participants will be asked to rate how stressful their day was the day before. The question is: "How stressful was your day yesterday?" The rating scale provided ranges from 1 (not at all) to 7 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Krafft, PhD, Principal Investigator — Mississippi State University
Locations (1):
- Mindfulness and Acceptance Processes Lab, Starkville, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share fully deidentified data sets. Any potentially identifying information including unusual demographics or combinations of demographics will be removed, but all other variables will be available to other researchers, journals or officials on reasonable request.
Supporting Information: Study Protocol
Time Frame: Within one year of the end of data collection, and remaining available indefinitely.
Access Criteria: There are no specific access criteria. The request must have a valid research-related purpose.

REFERENCES:
- [Background] Bangor, A., Kortum, P. T., & Miller, J. T. (2008). An empirical evaluation of the system usability scale. Intl. Journal of Human-Computer Interaction, 24(6), 574-594. https://doi.org/10.1080/10447310802205776
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Deci, E. L., & Ryan, R. M. (1985). The general causality orientations scale: Self-determination in personality. Journal of research in personality, 19(2), 109-134. https://doi.org/10.1016/0092-6566(85)90023-6
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Gregoire, S., Gagnon, J., Lachance, L., Shankland, R., Dionne, F., Kotsou, I., Monestès, J. L., Rolffs, J. L., & Rogge, R. D. (2020). Validation of the English and French versions of the multidimensional psychological flexibility inventory short form (MPFI-24). Journal of contextual behavioral science, 18, 99-110. https://doi.org/10.1016/j.jcbs.2020.06.004
- [Background] Guidelines for data processing and analysis of the IPAQ - short and long forms. (2005). IPAQ. https://sites.google.com/view/ipaq/score?authuser=0
- [Background] Hahn EA, Beaumont JL, Pilkonis PA, Garcia SF, Magasi S, DeWalt DA, Cella D. The PROMIS satisfaction with social participation measures demonstrated responsiveness in diverse clinical populations. J Clin Epidemiol. 2016 May;73:135-41. doi: 10.1016/j.jclinepi.2015.08.034. Epub 2016 Feb 27. PMID 26931288
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Health Measures. (2017). Global Health. http://www.healthmeasures.net/images/PROMIS/manuals/PROMIS_Global_Scoring_Manual.pdf
- [Background] Health Measures. (2014). Satisfaction With Social Roles and Activities. https://www.healthmeasures.net/images/promis/manuals/PROMIS_Satisfaction_with_Participation_in_Social_Roles_Scoring_Manual.pdf
- [Background] Kelley, M. L., Heffer, R. W., Gresham, F. M., & Elliott, S. N. (1989). Development of a modified treatment evaluation inventory. Journal of psychopathology and behavioral assessment, 11, 235-247.
- [Background] Knell G, Gabriel KP, Businelle MS, Shuval K, Wetter DW, Kendzor DE. Ecological Momentary Assessment of Physical Activity: Validation Study. J Med Internet Res. 2017 Jul 18;19(7):e253. doi: 10.2196/jmir.7602. PMID 28720556
- [Background] Krafft, J., Middleton, A., & Tadros, N. (2024). Is the Multidimensional Psychological Flexibility Inventory valid for ecological momentary assessment? A preliminary psychometric investigation. [Manuscript in preparation]. Department of Psychology, Mississippi State University
- [Background] Krafft, J., & Levin, M. E. (2021). Does the Cognitive Fusion Questionnaire measure more than frequency of negative thoughts?. Journal of Contextual Behavioral Science, 22, 63-67. https://doi.org/10.1016/j.jcbs.2021.09.002
- [Background] Markland, D., & Tobin, V. (2004). A modification to the behavioural regulation in exercise questionnaire to include an assessment of amotivation. Journal of Sport and Exercise Psychology, 26(2), 191-196. https://doi.org/10.1123/jsep.26.2.191
- [Background] Markland, D. (n. d.). Scoring the BREQ. http://exercise-motivation.bangor.ac.uk/breq/brqscore.php
- [Background] McLoughlin, S., Stapleton, A., & Hochard, K. D. (2022). Development and preliminary validation of the Value Clarity Questionnaire. PsyArXiv. https://doi.org/10.31234/osf.io/u97q3
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Rolffs JL, Rogge RD, Wilson KG. Disentangling Components of Flexibility via the Hexaflex Model: Development and Validation of the Multidimensional Psychological Flexibility Inventory (MPFI). Assessment. 2018 Jun;25(4):458-482. doi: 10.1177/1073191116645905. Epub 2016 May 5. PMID 27152011
- [Background] Wilson, P. M., Rodgers, W. M., Loitz, C. C., & Scime, G. (2006). It's Who I Am...Really! The Importance of Integrated Regulation in Exercise Contexts. Journal of Applied Biobehavioral Research, 11(2), 79-104. https://doi.org/10.1111/j.1751-9861.2006.tb00021.x
- [Background] Krafft, J., Klimczak, K. S., & Levin, M. E. (2022). Effects of cognitive restructuring and defusion for coping with difficult thoughts in a predominantly white female college student sample. Cognitive Therapy and Research, 46(1), 86-94.